CLINICAL TRIAL: NCT03767166
Title: A Prospective, Single Arm Study to Evaluate the Feasibility of the Archimedes Biodegradable Biliary and Pancreatic Stents Placement
Brief Title: The Archimedes Biodegradable Biliary and Pancreatic Stents
Acronym: ARCHIMEDES
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2275
Record Dates: First submitted 2018-11-20; First posted 2018-12-06 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Diseases
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Biodegradable biliary and pancreatic stents placement — Biodegradable biliary and pancreatic stents placement

SUMMARY:
This is a prospective, phase II, single-centre, non-randomised, single-arm study, enrolling patients with benign and malignant bilio-pancreatic diseases with an indication to biliary or pancreatic plastic stent positioning during ERCP.

On procedure day, the study team will confirm that the patient meets all the inclusion criteria and none of the exclusion criteria.

The patient will undergo the ABS insertion and monitored and follow-up accordingly to biodegration variant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication to position one ore more biliary plastic stents during ERCP
* Patients with an indication to position a pancreatic plastic stent during ERCP

Exclusion Criteria:

* Age < 18 y
* Life expectancy < 1 m,
* Inability to pass a guidewire through stricture
* Contra-indication for endoscopy or interventional radiology
* Presence of partial gastric resection
* Unsigned informing consent form, ICF
* Pregnancy
* Pseudo Klatskin tumors (metastases in the liver hilum) and gallbladder carcinoma

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with benign and malignant bilio-pancreatic diseases with an indication to biliary or pancreatic plastic stent positioning during ERCP.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Biodegradation time | 24 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderloni A, Fugazza A, Maroni L, Ormando V, Maselli R, Carrara S, Cappello A, Mangiavillano B, Omodei P, Preatoni P, Galtieri PA, Pellegatta G, Repici A. New biliary and pancreatic biodegradable stent placement: a single-center, prospective, pilot study (with video). Gastrointest Endosc. 2020 Aug;92(2):405-411. doi: 10.1016/j.gie.2020.02.049. Epub 2020 Mar 5. PMID 32145287